CLINICAL TRIAL: NCT02215837
Title: Randomized,Controlled,Multicenter Study of Autologous Tumor Lysate-pulsed Dendritic and Cytokine-induced Killer Cells(Ag-D-CIK) Combined With Chemotherapy for Gastric Cancer.
Brief Title: Study of Autologous Tumor Lysate-pulsed D-CIK Combined With Chemotherapy for Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shenzhen Hornetcorn Bio-technology Company, LTD (Industry)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Jingzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYK-Gastric Cancer
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2015-11

CONDITIONS: Gastric Cancer; Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases
Keywords: Gastric cancer; D-CIK; Autologous tumor lysate
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases | interventions — Drug Therapy; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy (Sham Comparator): After accepting chemotherapy according to NCCN guidelines, patients will just regularly follow up.
  Interventions: Drug: Chemotherapy
- Ag-D-CIK (Experimental): After accepting chemotherapy according to NCCN guidelines,patients will receive 3 cycles of autologous tumor lysate pulsed D-CIK treatment.
  Interventions: Drug: Chemotherapy; Biological: Ag-D-CIK

INTERVENTIONS:
Drug: Chemotherapy — Oxaliplatin 85mg/m2 IV over 2 hours, day 1; Leucovorin 400mg/m2 IV over 2 hours, day 1; 5-FU 400mg/m2 IV bolus on day 1, then 1200mg/m2/day for 2 days IV continuous infusion; Repeat every 2 weeks.
  Other Names: FOLFOX
Biological: Ag-D-CIK — 8×10^9 autologous tumor lysate pulsed D-CIK cells for each infusion, IV (in the vein) for 3 cycles, each cycle received four infusions on day 14, 16, 30 and 32.
  Arms: Ag-D-CIK

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of chemotherapy combined with autologous tumor Lysate-pulsed dendritic with cytokine-induced killer cell (Ag-D-CIK) for gastric cancer.

DETAILED DESCRIPTION:
40 patients with stage Ⅰ～Ⅲ Gastric Cancer,who had received surgery and kept their tumor tissue,will be randomly divided into group A（receive Ag-D-CIK treatment and chemotherapy) or group B（just receive chemotherapy),and the randomize ratio will be 1:1. Patients in group A will receive 3 cycles of Ag-D-CIK treatment (every 1 months) and 4 cycles of chemotherapy (every 2 weeks).Patients in group B will receive only 4 cycles chemotherapy（every 2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients who can accept curative operations
* 18~80 years old
* Histologically confirmed with gastric cancer at stage Ⅰ~Ⅲ
* Patients who can accept radical gastrectomy;
* Eastern Cooperative Oncology Group (ECOG) performance status was 0 - 1.

Exclusion Criteria:

* Hemoglobin<8.0 g/dL,White blood cell <3 x 10^9/L;Platelet count <75 x 10^9/L; ALT, AST, BUN and Cr more than normal limits on 3.0 times
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Pregnant or lactating patients
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV) or TreponemaPallidun (TP) infection
* Patients who are suffering from serious autoimmune disease
* Patients who had used long time or are using immunosuppressant
* Patients who had active infection
* Patients who are suffering from serious organ dysfunction
* Patients who are suffering from other cancer
* Other situations that the researchers considered unsuitable for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years
Quality of life (QOL) | 3 years
Phenotypic analysis of T cells | 1 years
  The number of CD3+ (or CD8+ or CD4+ or CD56+) T cell
Severity of adverse events | 1 years
  According to National Cancer Institute Common Terminology Criteria for Adverse Events（NCI-CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Hai Y Liu, Professor, Principal Investigator — Affiliated Tumor Hospital of Guangzhou Medical University immunotherapy center
Locations (2):
- China (2):
  - Affiliated Tumor Hospital of Guangzhou Medical University Immunotherapy center, Guangzhou, Guangdong
  - Jingzhou Central Hospital Immunotherapy center, Jingzhou, Hubei

IPD SHARING:
Plan to Share IPD: Undecided